CLINICAL TRIAL: NCT02828956
Title: Motivation to Change, Coping, and Self-Esteem in Adolescent Anorexia Nervosa
Status: Completed | Type: Observational
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: ANSOCQ_16
Record Dates: First submitted 2016-07-04; First posted 2016-07-12 (Estimated); Last update posted 2016-07-12 (Estimated); Status verified 2016-07

CONDITIONS: Personality Features in Anorexia Nervosa
Keywords: eating disorders; ANSOCQ; anorexia nervosa
MeSH Terms: conditions — Feeding and Eating Disorders; Anorexia Nervosa

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
By use of several questionaires, this study aimed at an investigation of the changes in motivation, symptoms, self-esteem and coping style in adolescent patients with anorexia nervosa.. The psychometric properties of the Anorexia Nervosa Stages of Change Questionnaire (ANSOCQ) and its relation to coping style and self-esteem were assessed. After a treatment period of nine months, clinical AN diagnosis and the body mass index (BMI) were re-assessed. Besides construct validity of the ANSOCQ, its predictive validity in terms of predicting the outcome of AN was assessed.

DETAILED DESCRIPTION:
N=92 adolescents referred to an eating disorders clinic meeting criteria for anorexia nervosa (AN) gave written informed consent to participate in this study and completed the ANSOCQ, the Eating Disorder Inventory (EDI-2), the Eating Attitudes Test (EAT), the Body Image Questionnaire (BIQ), two questionnaires measuring Self-Related Cognitions (SRC) and the Coping Across Situations Questionnaire (CASQ). After a treatment period of nine months, clinical AN diagnosis and the body mass index (BMI) were re-assessed. Exploratory factor analysis and logistic regressions were performed.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive cohort of patients aged 12-19 years with a certified diagnosis of anorexia nervosa

Exclusion Criteria:

* none

Ages: 12 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: N=92 adolescents referred to our eating disorders clinic meeting criteria for anorexia nervosa (AN).
Sampling Method: Non-Probability Sample
Enrollment: 92 (Actual)
Dates: Start 2010-01; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Stages of Change | 9 months
  The ANSOCQ measuring readiness to change in patients with anorexia nervosa.
Eating-Disorder inventory | 9 months
  91 item self-report measure assessing symptoms and attitudes related to eating disorders. It consists of 11 subscales (drive for thinness, bulimia, body dissatisfaction, effectiveness, interpersonal distrust, interoceptive awareness, asceticism, perfectionism, social insecurity, maturity fears and impulse regulation)
Rosenberg Self-esteem Scale | 9 months
  10 item self-report scale measure assessing self-esteem.
German Coping Across Situations Questionnaire | 9 months
  Questionnaire assessing coping behavior in four problem areas (school, parents, peers and the opposite sex). 20 items in each area.
Body Mass Index | 9 months
  Rating of weight in relation of a persons height
Body-Image-Questionnaire | 9 months
  A self-report measure assessing different aspects of body perception based on the model of semantic differentials.
Eating Attitudes Test | 9 months
  40 item self-report measure assessing eating attitudes and symptoms related to eating disorders. It consists of 3 subscales (dieting, bulimia and oral control).
Questionnaire for the assessment of dispositional self-awareness | 9 months
  Measure assessing private self-awareness (meta-cognitions regarding the private self) and public self-awareness (perception of oneself in presence of others).

CONTACTS AND LOCATIONS:
Overall Officials: Hans-Christoph Steinhausen, Principal Investigator — Department of Child and Adolescent Psychiatry and Psychotherapy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pauli D, Aebi M, Winkler Metzke C, Steinhausen HC. Motivation to change, coping, and self-esteem in adolescent anorexia nervosa: a validation study of the Anorexia Nervosa Stages of Change Questionnaire (ANSOCQ). J Eat Disord. 2017 Apr 17;5:11. doi: 10.1186/s40337-016-0125-z. eCollection 2017. PMID 28417002